CLINICAL TRIAL: NCT00312156
Title: Comparison of Efficacy and Safety of Insulin Detemir and NPH Insulin in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1379
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
The trial is conducted in Europe and Middle East. The aim of the trial is to compare the use of Insulin Detemir once or twice daily combined with mealtime Insulin Aspart against that of NPH Insulin once or twice daily combined with mealtime Insulin Aspart. The trial involves children and adolescents with Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Informed consent obtained
* BMI: 6-7 years: less than or equal to 19 kg/m2, 8-9 years: less than or equal to 20 kg/m2, 10-11 years: less than or equal to 22 kg/m2, 12-13 years: less than or equal to 24 kg/m2 and 14-17 years: less than or equal to 27 kg/m2.
* HbA1c equal to or less than 12.0%

Exclusion Criteria:

* Proliferate retinopathy or maculopathy
* Total daily insulin dose greater than 2.00 IU/kg
* Any condition or disease that rule out trial participation according to the judgement of the investigator.
* Mental incapacity, unwillingness or language barriers precluding understanding or cooperation.
* A life-style incompatible with trial participation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 2002-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks

SECONDARY OUTCOMES:
Adverse events
body weight
Antibodies
Blood glucose
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (42):
- Belgium (2):
  - Novo Nordisk Investigational Site, Bree
  - Novo Nordisk Investigational Site, Edegem
- Novo Nordisk Investigational Site, Rijeka, Croatia
- Denmark (4):
  - Novo Nordisk Investigational Site, Glostrup Municipality
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Viborg
- Finland (2):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Oulu
- France (4):
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Toulouse
- Germany (4):
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Kiel
  - Novo Nordisk Investigational Site, Stuttgart
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Petah Tikva, Israel
- Netherlands (3):
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Spijkenisse
  - Novo Nordisk Investigational Site, Utrecht
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Norway (4):
  - Novo Nordisk Investigational Site, Bodø
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Sarpsborg
  - Novo Nordisk Investigational Site, Tønsberg
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Spain (2):
  - Novo Nordisk Investigational Site, Leganés
  - Novo Nordisk Investigational Site, Madrid
- Sweden (6):
  - Novo Nordisk Investigational Site, Helsingborg
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
- Novo Nordisk Investigational Site, Zurich, Switzerland
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Stirling

REFERENCES:
- [Result] Robertson KJ, Schoenle E, Gucev Z, Mordhorst L, Gall MA, Ludvigsson J. Insulin detemir compared with NPH insulin in children and adolescents with Type 1 diabetes. Diabet Med. 2007 Jan;24(1):27-34. doi: 10.1111/j.1464-5491.2007.02024.x. PMID 17227321
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com